CLINICAL TRIAL: NCT06540118
Title: Food Is Medicine for Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Cheryl A. Anderson, MPH, PhD, Professor and Dean, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24RPGFIM1198191
Record Dates: First submitted 2024-07-24; First posted 2024-08-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Heart Failure，Congestive; Heart Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — myotubularin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: By the nature of the dietary intervention, it is impossible to blind participants to study arm assignment. However, research staff collecting outcome data, apart from dietary adherence data, will remain blinded to participants' assigned study arm throughout data collection. Additionally, the statistician(s) analyzing data for efficacy of the intervention will use a dataset with study arm masked in order to remain blinded to the assigned intervention for the final analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 Medically Tailored Meals (MTM) + snacks (Experimental): Participants will receive 15 medically tailored meals (MTM) per week, plus snacks, for 12 weeks.
  Interventions: Other: 15 Medically Tailored Meals (MTM) per week
- 14 Medically Tailored Meals (MTM) (Experimental): Participants will receive 14 medically tailored meals (MTM) per week for 12 weeks.
  Interventions: Other: 14 Medically Tailored Meals (MTM) per week

INTERVENTIONS:
Other: 15 Medically Tailored Meals (MTM) per week — 15 heart-healthy medically tailored meals delivered to participants each week. Meals include breakfast, lunch, dinner, and snack to consume Monday-Friday.
  Arms: 15 Medically Tailored Meals (MTM) + snacks
Other: 14 Medically Tailored Meals (MTM) per week — 14 heart-healthy medically tailored meals delivered to participants each week. Meals include lunch and dinner to consume Monday-Sunday.
  Arms: 14 Medically Tailored Meals (MTM)

SUMMARY:
This study will look at the effects of providing medically tailored meals (MTMs) to people with heart disease for twelve weeks. The primary outcome of the study is the quality of the diet being consumed in week 12 of the study, as determined by the "Healthy Eating Index."

DETAILED DESCRIPTION:
This study will look at the effects of providing medically tailored meals (MTMs) to people with heart disease for twelve weeks. Sixty adults with heart failure will be recruited from the San Diego and San Francisco Bay Area of California. They will be randomly assigned to two groups: 1) a group that receives 15 "medically tailored meals" plus snacks each week for 12 weeks, 2) a group that receives 14 "medically tailored meals" each week for 12 weeks. The primary outcome of the study is the quality of the diet being consumed in week 12 of the study, as determined by the "Healthy Eating Index". Many other secondary outcomes will be assessed including both qualitative factors (e.g., satisfaction, preferences, adherence) and quantitative clinically measures (e.g., blood cholesterol, blood pressure, weight).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study
* Living in San Diego or the Bay Area of California
* Reported congestive heart failure (CHF) diagnosis
* Current diet can be improved
* Willing to eat all meals provided by the study

Exclusion Criteria:

* Diagnosed with end-stage heart failure
* Diagnosed with diabetes (type 1 or uncontrolled type 2)
* Currently taking insulin and/or meglitinides medications
* Currently taking Glucagon-Like Peptide-1 (GLP-1) Agonists medications and not stable on a maximum maintenance dose for a minimum of 1 month
* Hemoglobin A1c (HbA1c) results >8 %
* Life expectancy of <1 year
* Pregnancy or lactation
* Known severe allergic reactions and/or food intolerances that would interfere with the ability to eat study-provided meals, including foods that are prepared in a facility that works with the allergen
* Current smoker or tobacco use within the past year
* Planning to leave San Diego or the Bay Area during the course of the study
* Unable to communicate reasonably well either orally or through written material in English
* Those who, in the opinion of the investigators, cannot reliably complete the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Change in diet quality at Week 12, as determined by the Healthy Eating Index (HEI) | Baseline and Week 12
  HEI will be used to determine diet quality based on dietary recall data collected via Nutrition Data System for Research (NDSR) software. HEI scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations and dietary patterns published in the Dietary Guidelines for Americans.

SECONDARY OUTCOMES:
Participant satisfaction with delivery of medically tailored meals for individuals with heart failure | Week 4 and Week 12
  Participant satisfaction will be assessed using a study-specific self-administered questionnaire that uses a 5-point Likert scale. Participants will be asked to rate their experiences with multiple aspects of the provided study meals (including taste, variety, quality, cultural appropriateness, amount of food, visual appeal, and delivery) from "poor" to "excellent".
Dietary adherence to meal assignment using daily food diaries and 24-hour dietary recalls | Baseline and Weeks 4, 6, 8, and 12
  Participants' qualitative daily food diaries and quantitative dietary analyses based on interviewer-assisted dietary recalls using Nutrition Data System for Research (NDSR) software will be combined to determine the proportion of provided meals that participants consumed.
Change in reported access to healthy foods as assessed by the Food Consumption Score (FCS) | Baseline, Week 12, and Week 24
  The Food Consumption Score aggregates household-level data on the diversity and frequency of food groups consumed over the previous seven days, which is then weighted according to the relative nutritional value of the consumed food groups. The Food Consumption Score scale ranges from 0-112, with higher scores indicating better food consumption status.
Change in reported food security as assessed by the Food Insecurity Experience Scale (FIES) | Baseline, Week 12, Week 24
  The Food Insecurity Experience Scale (FIES) consists of eight questions regarding people's access to adequate food during the last 30 days. The raw score scale ranges from 0-8, with a higher score indicating more food insecurity experiences. Scale items are analyzed together as a scale, not be reported in terms of percent of positive responses to individual questions. The classifications of food insecurity severity based on responses may be described as mild, moderate, and severe food insecurity.
Change in reported food security as assessed by the Short Form of the U.S. Adult Food Security Survey Module | Baseline, Week 12, Week 24
  The 6-item survey collects information about whether participants had access to and were able to afford enough food in the last 30 days. The survey allows for stratification of participants into one of four food security categories based on their responses - high food security, marginal food security, low food security, and very low food security. The raw score scale ranges from 0 - 6, with a higher score indicating lower food security.
Change in mean blood pressure | Baseline and Week 12
  Mean blood pressure will be calculated based on 3 consecutive readings in the research clinic during each in-person study visit.
Change in blood lipid levels | Baseline and Week 12
Change in Hemoglobin A1C (HbA1C) levels | Baseline and Week 12
Change in weight | Baseline and Week 12
  Weight will be measured by study personnel at each in-person study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Anderson, PhD, MPH, MS, Principal Investigator — UC San Diego; Christopher Gardner, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No